CLINICAL TRIAL: NCT00507156
Title: Postconditioning Used to Limit Final Infarct Size in Patients With Acute ST-segment Elevation Myocardial Infarction
Brief Title: Postconditioning in the Treatment of Acute ST-segment Elevation Myocardial Infarction
Acronym: POSTCON
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Thomas Engstrom, Chief Consultant, Rigshospitalet, Denmark
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KF 01 326257
Record Dates: First submitted 2007-07-23; First posted 2007-07-25 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: ST-segment Myocardial Infarction

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Mek postcon (Experimental): Re-opening of the infarcted coronary artery by several balloon inflations separated by reperfusion of the vessel.
  Interventions: Procedure: Mechanical postconditioning
- Standard treatment (Active Comparator): Standard treatment (primary PCI)
  Interventions: Procedure: Standard primary PCI

INTERVENTIONS:
Procedure: Standard primary PCI — Acute re-opening of the occluded coronary artery
  Arms: Standard treatment
Procedure: Mechanical postconditioning — Mechanical postconditioning with 4 cycles 30/30 sek balloon inflations
  Arms: Mek postcon

SUMMARY:
Standard treatment of patients with acute ST-segment elevation myocardial infarction consist of acute re-opening of the occluded coronary artery (primary PCI). Despite successful treatment of the epicardial vessel reperfusion is sometimes inadequate leading to large final infarct sizes. This phenomenon is known as the reperfusion injury. Several animal studies have indicated that graded re-opening of the artery may limit tissue damage. Generally this is referred to as mechanical postconditioning.

The study investigates the effect on final infarct size evaluated by magnetic resonance scan of postconditioning of ST-segment elevation myocardial infarctions. Mechanical postconditioning is performed by means of several balloon inflations in the injured vessel following its acute re-opening.

DETAILED DESCRIPTION:
Please see above

ELIGIBILITY:
Inclusion Criteria:

* Patients more than 18 years
* STEMI < 12 hours
* TIMI 0-1 in infarct related artery

Exclusion Criteria:

* Multivessel disease (stenoses in non-infarct related arteries >70%)
* Cardiogenic shock
* Left main occlusions
* Lesions that cannot be treated with stents
* Previous CABG
* Pregnancy
* Severe renal insufficiency
* Previous extensive Q-wave infarction
* LBBB

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-07; Primary Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
Final infarct size evaluated by MR | 3 month

SECONDARY OUTCOMES:
MACE (death, re-infarction, TLR) | 1, 15 month
Stent thrombosis | 15 month

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Engstrom, D.Sci., PhD, Study Chair — Cheif Consultant
Locations (1):
- Cardiac Catherization Lab., Heart Center, Rigshospitalet, University of Copenhagen, Copenhagen, Denmark

REFERENCES:
- [Derived] Lonborg J, Holmvang L, Kelbaek H, Vejlstrup N, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Treiman M, Jensen JS, Engstrom T. ST-Segment resolution and clinical outcome with ischemic postconditioning and comparison to magnetic resonance. Am Heart J. 2010 Dec;160(6):1085-91. doi: 10.1016/j.ahj.2010.09.026. PMID 21146662
- [Derived] Lonborg J, Kelbaek H, Vejlstrup N, Jorgensen E, Helqvist S, Saunamaki K, Clemmensen P, Holmvang L, Treiman M, Jensen JS, Engstrom T. Cardioprotective effects of ischemic postconditioning in patients treated with primary percutaneous coronary intervention, evaluated by magnetic resonance. Circ Cardiovasc Interv. 2010 Feb 1;3(1):34-41. doi: 10.1161/CIRCINTERVENTIONS.109.905521. Epub 2010 Jan 26. PMID 20118154